CLINICAL TRIAL: NCT06630858
Title: Comparison of The Effects of Subcostal Anterior Quadratus Lumborum Block and Intrathecal Morphine on Postoperative Acute Pain in Laparoscopic Nephrectomy Surgery: A Randomized, Single-Blind, Non-Inferiority Trial
Brief Title: Intrathecal Morphine vs. Quadratus Lumborum Block for Pain in Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Professor Dr, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: S-QLBITMLSN
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Analgesia; Acute Pain; Patient Controlled Analgesia
Keywords: Subcostal Anterior Quadratus Lumborum Block; Laparoscopic nephrectomy; Intrathecal morphine
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program;Research Randomizer (Urbaniak and Plous 2013).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based;Research Randomizer; (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio.
  A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist who will administer the block/blocks about which group the patient is in immediately before administration. Researchers, patients, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S-QLB3 (Active Comparator): S-QLB3 block (0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline) + iv morphine-PCA
  Interventions: Procedure: Subcostal Anterior Quadratus Lumborum Block; Drug: Patient Controlled Analgesia (IV PCA)
- Group ITM (Active Comparator): ITM Morphine (a total of 0.2 mg of morphine sulfate + 7.5 mg isobaric (plain) bupivacaine ) + iv morphine-PCA
  Interventions: Procedure: Intrathecal Morphine; Drug: Patient Controlled Analgesia (IV PCA)

INTERVENTIONS:
Procedure: Subcostal Anterior Quadratus Lumborum Block — S-QLB3 block will be performed 30 min. before general anesthesia. For anterior QL block via subcostal approach, 0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline will be injected into the interfacial plane between the QLM and PMM.
  Arms: Group S-QLB3
Procedure: Intrathecal Morphine — Intrathecal morphine will be performed (a total of 0.2 mg of morphine sulfate + 7.5 mg isobaric bupivacaine).
  Arms: Group ITM
Drug: Patient Controlled Analgesia (IV PCA) — IV morphine-PCA will be applied postoperatively for 24 hours . IV-PCA: The requested dose will be 1mg morphine, the lock-in time will be 6 minutes, the 4-hour limit will be 20 mg morphine.

SUMMARY:
In this study, it was aimed to evaluate the effects of subcostal anterior quadratus lumborum block (S-QLB3) and İntrathecal morphine (ITM) on postoperative acute pain scores and opioid consumption in the first 24 hours after laparoscopic nephrectomy surgery.

DETAILED DESCRIPTION:
For all patients undergoing surgery, analgesic medications and techniques are routinely administered preoperatively, intraoperatively, and postoperatively to relieve their pain. Depending on the method applied, patients' analgesic needs in the recovery room and ward after surgery may vary. In patients undergoing laparoscopic nephrectomy, multimodal analgesia (paracetamol, nonsteroidal anti-inflammatory drugs, and opioids) is routinely applied in our clinic, utilizing various regional techniques or intravenous analgesics .

Opioids are the gold standard for postoperative pain control; however, they increase the incidence of opioid-related adverse effects such as dizziness, nausea, vomiting, constipation, and respiratory depression. Therefore, minimizing opioid use and its side effects is essential for postoperative pain control. Regional analgesia is a beneficial method for reducing opioid consumption and postoperative pain. It may also reduce postoperative morbidity and mortality.

Recently, interfascial plane blocks have been used for postoperative pain control in abdominal surgeries. The quadratus lumborum block (QLB) is a relatively new interfascial plane block technique in which local anesthetics are injected adjacent to the quadratus lumborum muscle. There are four different approaches to the QLB: anterior, intramuscular, lateral, and posterior. Anterior QLB involves the injection of a local anesthetic between the quadratus lumborum (QL) muscle and the psoas muscle. The dermatome coverage is determined by the injection site. The injection of local anesthetic anterior to the QL muscle potentially allows the drug to spread into the thoracic paravertebral space, blocking the somatic and sympathetic nerves of the lower thoracic segments. This situation helps us achieve more effective analgesia in abdominal surgeries.

Intrathecal morphine (ITM) is an emerging strategy for postoperative analgesia following major abdominal surgery. Traditional spinal analgesia protocols often rely on continuous thoracic epidural anesthesia due to their ability to provide adequate analgesia with a few cardiopulmonary complications. However, epidural anesthesia is also associated with more frequent perioperative hypotension, technical failures, increased fluid administration, and longer length of stay (LOS). Therefore, ITM is an attractive alternative because it offers easier administration, potent efficacy at low doses, and reduced postoperative complications, providing a form of spinal analgesia that can be used when epidural catheters are contraindicated.

The analgesic properties of ITM have been demonstrated in recent studies involving cardiac, gynecological, spinal, orthopedic, urological, colorectal, hepatopancreatobiliary, and major abdominal surgeries. With an estimated duration of action of up to 24 hours, these studies have focused on the initial postoperative recovery period and generally found lower pain scores and, in some cases, reduced early postoperative opioid requirements. Intrathecal morphine has been successfully used for postoperative pain in various surgeries. Being a hydrophilic opioid, morphine's limited sequestration in adipose tissue delays its clearance from the cerebrospinal fluid compared to other opioids. As a result, the analgesic effects of intrathecal morphine last longer, providing up to 24 hours of analgesia without the need for indwelling catheters or continuous infusions. Direct injection into the intrathecal space also allows morphine to act directly on opioid receptors in the brain and the substantia gelatinosa of the spinal cord, providing a potent analgesic response.

In this study, it was aimed to determine whether the subcostal anterior quadratus lumborum block (S-QLB3) is non-inferior to intrathecal morphine (ITM) in terms of postoperative 24-hour opioid consumption in patients undergoing laparoscopic nephrectomy.

The H0 hypothesis of study is that the mean difference in postoperative 24-hour morphine consumption between S-QLB3 and ITM is less than or equal to the non-inferiority margin.

Patients will be divided into two groups:

Group S-QLB3:A unilateral S-QLB3 block will be performed (0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline). In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

Group ITM: Intrathecal morphine will be performed (5 mcg/kg preservative-free morphine (maximum 200 mcg) + 7.5 mg isobaric bupivacaine). In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years who had an American Society of Anesthesiologists (ASA) Physical Status classification I-III

Exclusion Criteria:

* refusal to participate in the study
* body mass index>35 kg/m2
* contraindications to peripheral nerve blocks or spinal anesthesia (e.g., the presence of coagulopathy or pre-existing local or systemic infection etc.)
* unable to perform regional anesthesia because of anatomical deformity
* clinically important cardiovascular and cerebrovascular diseases or preexisting significant organ dysfunction (eg, hepatic, renal or respiratory disorders)
* allergic reaction to any study drugs
* history of substance
* abuse within the three-month period prior to surgery, chronic opioid use for at least a continuous administration of opioids for a duration of 30 days at daily morphine-equivalent dose ≥15 mg/d (1)
* psychiatric illness and disorder in communication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cumulative equivalent morphine consumption in the first 24 hours after surgery | postoperative day 1
  Cumulative equivalent morphine consumption in the first 24 hours after surgery will be measured. Patients can request opioids via a PCA device when their NRS score is ≥4. In cases where rescue analgesia is required (NRS score ≥4), 25 mg IV meperidine was administered in the recovery unit, and 50 mg IM meperidine was administered in the ward.

SECONDARY OUTCOMES:
Postoperative pain scores | postoperative day 1
  Pain status at rest and while activity will be assessed by NRS score at 0, 3, 6, 12, and 24 hours after surgery. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Patients satisfaction and quality of pain management | preoperatively, postoperative day 1 and the 1 day of discharge
  Patientsmanagement satisfaction and quality will be evaluated using the Turkish version of the 15-item quality of recovery (QoR-15) scale (1,2). The QoR-15 is measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale is a patient-perceived, well-validated, global outcome measure of postoperative recovery, and provides an aggregate score ranging from 0 (extremely poor recovery) to 150 (excellent recovery).
intraoperative total remifentanil consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes.
  The total amount of remifentanil consumed will be recorded.
The heart rate measurement | The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes
  The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.
The mean arterial pressure measurement | The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes.
  The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.
The number of patients requiring rescue analgesics | postoperative day 1
  The number of patients requiring rescue analgesics will be recorded over 24 hours.
Cumulative equivalent morphine consumption in the first 12 hours after surgery | postoperative day 1
  Cumulative equivalent morphine consumption in the first 12 hours after surgery will be measured. Patients can request opioids via a PCA device when their NRS score is ≥4 and 25 mg IV meperidine was administered in the recovery unit, and 50 mg IM meperidine was administered in the ward.
The number of patients requiring postoperative antiemetics. | postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, and 24 hours after extubation. For PONV prophylaxis, patients will be routinely administered 8 mg IV dexamethasone before induction and 0.15 mg/kg (IVA) IV ondansetron 20 minutes before the end of the procedure. If a score of 3 or more is recorded, 4 mg IV ondansetron will be administered and repeated after 4 hours if required. Despite the administration of ondansetron, if the score is ≥3, the patients will be administered 10 mg IV metoclopramide diluted in 100 ml saline solution as an IV infusion. The number of patients who receive antiemetic treatment will be recorded. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
Sedation score | postoperative day 1
  Sedation score will be assessed at 0, 3, 6, 12, and 24 hours after extubation. (0: awake, 1: drowsy but easily arousable, 2: very drowsy but still arousable, 3: difficult to rouse)
Time of first analgesic request | postoperative day 1
  Time at which the first analgesic is requested
The morbidity of patients | Postoperative 1 month on an average
  The patients comorbidities will be assessed using the Charlson Comorbidity Index.
Complications | Postoperative 1 month on an average
  The following complications observed until discharge (30 days) will be recorded: post-dural puncture headache, respiratory depression, nausea, vomiting, itching, sedation, nerve injury, hematoma or infection at the puncture site, visceral organ injury, pneumothorax, retroperitoneal hematoma, quadriceps weakness, and LAST. The severity of observed complications will be assessed using the Clavien-Dindo classification. Additionally, the Comprehensive Complication Index will be used to evaluate the patients overall postoperative morbidity.
The incidences of post-operative pruritus | Postoperative day 1
  The presence and severity of pruritus will be assessed using a four-point scale where 0 indicates no pruritus, 1 indicates mild pruritus, 2 indicates moderate pruritus, and 3 indicates severe pruritus. A score of ≥1 will be considered the presence of pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Kaya, MD, Principal Investigator — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayis University, Samsun
  - OndokuzMAyis University, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaya C, Dost B, Turunc E, Ustun YB, Kibar AN, Cebeci H, De Cassai A, Elsharkawy H. Unilateral subcostal anterior quadratus lumborum block versus intrathecal morphine for postoperative pain in laparoscopic nephrectomy: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jul 10:rapm-2025-106844. doi: 10.1136/rapm-2025-106844. Online ahead of print. PMID 40639953